CLINICAL TRIAL: NCT02315846
Title: Role of Acetylcholinesterase for the Diagnosis of Postoperative Delirium in Patients Needing Postoperative Monitoring
Brief Title: Acetylcholinesterase in Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Christoph Schramm, M.D., Principal Investigator, Heidelberg University
Other Study IDs: S452/2013
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood-serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The level of acetylcholinesterase is suspected to correlate with postoperative delirium. The investigators therefore score patients once preoperatively and twice postoperatively with the german version of the delirium-score NuDESC (Nursing Delirium Screening Scale) and compare the results with the acetylcholinesterase activity, butyrylcholinesterase activity and the serum anticholinergic activity (SAA) at corresponding time points.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Elective surgery

Exclusion Criteria:

* Preexisting psychiatric or neurological disease
* No surgery
* Reduced level of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients in the head clinic of the University of Heidelberg, Germany with surgery, that requires them to stay in Hospital for at least 3 days postoperatively
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change of acetylcholinesterase (U/l) | one day before surgery, 1-24h after surgery, 25-72h after surgery
  change of acetylcholinesterase in units per litre

SECONDARY OUTCOMES:
change of NuDESC | one day before surgery, 1-24h after surgery, 25-72h after surgery
  change of nursing delirium screening score
change of medication | one day before surgery, 1-24h after surgery, 25-72h after surgery
  change of medication, that could influence a delirium
ICD-codes of main disease | 25-72h after surgery
  International classification of diseases-code of main disease
ICD-codes of coexisting diseases | 25-72h after surgery
  International classification of diseases-codes of coexisting diseases

CONTACTS AND LOCATIONS:
Overall Officials: Konstanze Plaschke, PhD, Study Director — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany